CLINICAL TRIAL: NCT06893887
Title: Exploratory Cohort Study and Mechanistic Research on Individualized Comprehensive Treatment After Standard Treatment for Advanced Hepatocellular Carcinoma
Brief Title: Individualized Comprehensive Treatment for Advanced Hepatocellular Carcinoma
Acronym: ICT-HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Tianyinshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2025-KT-005-01
Record Dates: First submitted 2025-02-27; First posted 2025-03-25 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma(HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; apatinib; icaritin; SHR-1701; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Arm 1 (Experimental): XELOX/FOLFOX4+ Adebelizumab + Apatinib+Icaritin
  Interventions: Drug: FOLFOX4; Drug: Adebrelimab
- Arm 2 (Experimental): Adebelizumab + Apatinib+Icaritin
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Drug: Icaritin
- Arm 3 (Experimental): SHR1701+ Apatinib+Icaritin
  Interventions: Drug: Apatinib; Drug: Icaritin; Drug: SHR-1701
- Arm 4 (Experimental): QL1706+ Apatinib+Icaritin
  Interventions: Drug: Apatinib; Drug: Icaritin; Drug: QL1706
- Arm 5 (Experimental): The original targeted combination immunotherapy+HAIC
  Interventions: Procedure: HAIC; Drug: The original treatment regimen
- Arm 6 (Experimental): SHR1701+ Apatinib+Icaritin，intrahepatic progression
  Interventions: Drug: Apatinib; Drug: Icaritin; Drug: SHR-1701
- Arm 7 (Experimental): QL1706+ Apatinib+Icaritin，extrahepatic progression
  Interventions: Drug: Apatinib; Drug: Icaritin; Drug: QL1706
- Arm 8 (Experimental): SHR1701+Bevacizumab+Icaritin
  Interventions: Drug: Icaritin; Drug: SHR-1701; Drug: Bevacizumab
- Arm 9 (Experimental): QL1706+Bevacizumab+Icaritin
  Interventions: Drug: Icaritin; Drug: QL1706; Drug: Bevacizumab
- Arm 10 (Experimental): Local treatment of oligometastases (such as radiotherapy, RFA, etc.) + the original targeted and immunotherapy.
  Interventions: Procedure: Local treatment; Drug: The original treatment regimen

INTERVENTIONS:
Drug: FOLFOX4 — FOLFOX4 was administered by oxaliplatin 85 mg/m² d1+ leucovorin 200 mg/m² d1-2+ fluorouracil 400 mg/m² 2 h→ 600 mg/m² 24 h d1-2 q2w, with a total of 4 cycles
  Arms: Arm 1
Drug: Adebrelimab — Adebrelimab 1200mg, intravenous infusion, every 3 weeks
  Arms: Arm 1; Arm 2
Drug: Apatinib — Apatinib 250mg, oral, once daily.
  Arms: Arm 2; Arm 3; Arm 4; Arm 6; Arm 7
Drug: Icaritin — Epimedium extract soft capsules 2.4g, oral, 2 times daily.
  Arms: Arm 2; Arm 3; Arm 4; Arm 6; Arm 7; Arm 8; Arm 9
Drug: SHR-1701 — SHR1701，30mg/kg, intravenous infusion, every 3 weeks, use for up to 2 years at most.
  Arms: Arm 3; Arm 6; Arm 8
Drug: QL1706 — QL1706，5mg/kg, intravenous infusion, every 3 weeks, use for up to 2 years at most.
  Arms: Arm 4; Arm 7; Arm 9
Drug: Bevacizumab — Bevacizumab 7.5mg, intravenous infusion, once every 3 weeks.
  Arms: Arm 8; Arm 9
Procedure: HAIC — Hepatic Arterial Infusion Chemotherapy
  Arms: Arm 5
Procedure: Local treatment — Local treatment of oligo-metastases.
  Arms: Arm 10
Drug: The original treatment regimen — Continue the original targeted therapy combined with immunotherapy. dosage, dosage form,frequency of administration was the same as before.
  Arms: Arm 10; Arm 5

SUMMARY:
This project is a prospective, multi-center, multi-cohort exploratory clinical study. It focuses on patients with advanced hepatocellular carcinoma who experience disease progression after first-line standard therapy. Based on different patterns of disease progression, patients will receive relevant systemic treatments, either with or without local interventional therapy. The primary endpoint is progression-free survival (PFS), while secondary endpoints include overall survival (OS), 1-year OS rate, objective response rate (ORR), disease control rate (DCR), duration of remission (DOR), and safety. Additionally, the study will explore the correlation between patients' clinical pathological characteristics, serum biomarkers, and clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female
2. Hepatocellular carcinoma patients diagnosed by cytology or tissue puncture, or who meet clinical diagnostic criteria and cannot be treated with radical treatment (radical surgery, ablation, radiotherapy, etc.)
3. Disease progression after first-line targeted combined immune system therapy (as per RECIST1.1 criteria)
4. Life expectancy exceeds 3 months
5. ECOG physical condition score 0~1
6. Women of childbearing age must have a serum pregnancy study done within 7 days before the first medication, and the result is negative. Female subjects of reproductive age and male subjects whose partners are women of reproductive age must consent to contraception within 24 weeks from the date of signing the informed consent to the last administration of the study drug
7. Before the first dose of the investigational drug, the laboratory test values met the following conditions: ①blood routine (no blood transfusion within 14 days before screening, no hematopoietic stimulating drug correction) : white blood cell count (WBC) ≥ 2.0 × 109/L; platelet (PLT) ≥ 60× 109/L; hemoglobin content (HGB) ≥ 8.0 g/dL; ② Liver function: aspartate transferase (AST) ≤ 2.5x ULN; alanine aminotransferase (ALT) ≤ 2.5 x ULN; Serum total bilirubin (TBIL) ≤ 1.5 x ULN (except Gilbert syndrome total bilirubin ≤ 3.0 mg/dL); ③ Renal function: serum creatinine ≤ 1.5 x ULN or creatinine clearance rate (CrCl) ≥ 50 mL/minute; ④ Coagulation function: international normalized ratio (INR) ≤ 1.5 x ULN, activated partial thromboplastin time (APTT) ≤ 1.5 x ULN (only for patients who are not currently receiving anticoagulant therapy, patients who are currently receiving anticoagulant therapy should receive a steady dose of anticoagulant therapy)
8. The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with the follow-up

Exclusion Criteria:

1. Pathological types of other non-hepatocellular carcinomas, including fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc. previously confirmed by histology/cytology
2. Child-Pugh grade of liver function ≥7 points
3. Major cardiovascular impairment in the 6 months prior to initial administration of the drug, such as a New York Heart Association (NYHA) Class II or higher history of congestive heart failure, unstable angina, myocardial infarction or stroke, or arrhythmia associated with hemodynamic instability; Corrected QT (QTc) interval lengthening >480ms
4. Other malignancies developed ≤ 5 years before the first dose, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery (hormone therapy for non-metastatic prostate cancer or breast cancer is allowed)
5. Have had an active autoimmune disease in the past 2 years that requires systemic treatment, including but not limited to autoimmune hepatitis, lupus erythematosus, etc
6. Uncontrolled active infection, such as active tuberculosis, HIV infection, etc.; Patients with HBV-DNA replication level below 10000IU/mL and continuous oral antiviral therapy could be enrolled.
7. Had undergone major surgery in the 28 days prior to randomization or planned to undergo major surgery during the study period
8. Use of live attenuated vaccine within 28 days prior to randomization, or anticipated use of such live attenuated vaccine during the study period (patients are not allowed to receive live attenuated influenza vaccine 4 weeks prior to randomization, during treatment, and within 5 months after the final administration of adbelizumab)
9. Received any other investigational drug treatment or participated in another interventional clinical study within 4 weeks prior to signing the ICF
10. Use of corticosteroids (> 10 mg/ day prednisone or equivalent dose) or other immunosuppressants within ≤ 14 days prior to the first dose of the study drug. Allowing inhaled or topical use of steroids and adrenal replacement steroids in the absence of active autoimmune disease; Patients received systemic immunosuppressive drugs (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] drugs) within 1 week prior to randomization. Patients receiving short-term, systemic immunosuppressant therapy, such as glucocorticoids for nausea, vomiting, or anaphylaxis management or prevention, may be enrolled in the study after investigator review. To allow the use of inhaled corticosteroids in patients with chronic obstructive pulmonary disease, corticosteroids such as fluhydrocortisone in patients with postural hypotension, and low-dose glucocorticoid supplements for adrenal insufficiency; Known mental illness, alcoholism, inability to quit smoking, drug or substance abuse
11. In the investigator's judgment, the subjects have other factors that may lead to the forced termination of the study, such as non-compliance with the protocol, other serious illnesses (including mental illness) requiring combined treatment, serious laboratory abnormalities, family or social factors that may affect the safety of the subjects, or the collection of data and samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
PFS（Progression-free Survival） | 24 months
  Progression-free survival (PFS) was defined as the time from treatment initiation on Day 1 to the earliest occurrence of radiologically confirmed disease progression, as assessed by tumor imaging, or death from any cause, whichever came first. Evaluations were conducted by the investigator in accordance with RECIST v1.1.

SECONDARY OUTCOMES:
OS(Overall survival) | 48 months
  Overall survival (OS) was defined as the duration from treatment initiation on Day 1 to death from any cause.
ORR(Objective response rate) | 24 months
  Objective response rate (ORR) was defined as the proportion of subjects achieving a complete response (CR) or partial response (PR), as assessed by the investigator according to RECIST v1.1, from the initiation of treatment on Day 1.
DCR(Disease control rate ) | 24 months
  Disease control rate (DCR) was defined as the proportion of subjects achieving a complete response (CR), partial response (PR), or stable disease (SD) lasting ≥8 weeks, as assessed by the investigator according to RECIST v1.1, from the initiation of treatment on Day 1.
DOR(Duration of Response) | 24 months
  Duration of response (DOR) was defined as the time from the first documented objective response (CR or PR) to the earliest occurrence of radiological disease progression or death from any cause, whichever occurred first. Both response and progression were evaluated by the investigator according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- China Pharmaceutical University Affiliated Nanjing Tianyinshan Hospital, Nanjing, Jiangsu, China